CLINICAL TRIAL: NCT01674452
Title: Home-based Exercises for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Maria Elisa Pimentel Piemonte, PT; PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPNEC003
Record Dates: First submitted 2012-08-13; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Cerebrovascular Disorders; Brain Infarction; Brain Ischemia; Stroke
Keywords: Stroke; Exercise and Physical Fitness
MeSH Terms: conditions — Cerebrovascular Disorders; Brain Infarction; Brain Ischemia; Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- home-based group (Experimental)
  Interventions: Behavioral: home-based group (HBG)
- supervised exercise group (Active Comparator)
  Interventions: Behavioral: supervised exercise group (SEG)
- control (No Intervention): Control group:no intervention

INTERVENTIONS:
Behavioral: home-based group (HBG) — Participants in the home-based group (HBG) were advised to exercise, a minimum of 4 times per week, but they were encouraged to exercise a total of 5-7 days per week. After individual assessment, a group of home-exercise selected of the manual was explained and performed one by one. The home-exercises were re-executed at each fortnightly visit, when necessary corrections were made and the next step stipulated by manual was taken, according to the patient's progress.
  Other Names: Home-based exercise supported by an illustrated manual
  Arms: home-based group
Behavioral: supervised exercise group (SEG) — Patients in the supervised exercise training group (SEG) participated in supervised individual exercise sessions 2 times per week. A physical therapist supervised these sessions. Exercise sessions included: 30 minutes of global exercises that involved stretching, range of motion, muscle strengthen and another 30 minutes of functional training (gait, balance and use of the arm in daily activities).
  Other Names: Conventional supervised exercise training
  Arms: supervised exercise group

SUMMARY:
The aim of this study is the development and the implementation of a new protocol about home-based exercises, supported by an illustrated manual, for the treatment of individuals with stroke.

The hypothesis is that this group of patients who are going to carry out the training of this study protocol are going to show improvement in measured parameters (functionality and physical performance), which allows this protocol to be improved and published as a proposal of physiotherapeutic treatment.

DETAILED DESCRIPTION:
1. Program Development: 27 exercises were selected, based on the most frequent motor alterations present in hemiparesis. Three modes were created for each exercise: assisted active, active and resisted active executions. Besides explanatory text, there were illustrative photos for all exercises and their modes.
2. Program Execution: All groups were submitted to a motor evaluation utilizing the Fugl-Meyer Assessment (FMA) and functional evaluation utilizing the Functional independence measure (FIM). After assessment, for the patients of the home-based exercise group (HBG) a group of home exercises was selected for each patient; these exercises were explained and performed one by one. The home-exercises were re-executed at each fortnightly visit, when any necessary correction was made. The next steps stipulated by the manual were taken, providing the patients with more complex exercises according to their progress. The patients in the supervised exercise training group (SEG) participated in supervised individual exercise sessions two times per week. A physical therapist supervised these sessions. Exercise sessions included: 30 minutes of global exercises that involved stretching, range of motion, muscle strengthen and another 30 minutes of functional training (gait, balance and use of the arm in daily activities).The control group (CG) was assessed but reluctant or unable to regularly attend a supervised exercise program. The groups were reassessed after six months.
3. Program assessment: The Fugl-Meyer Assessment score and the Functional independence measure score, measured at baseline and after six months, were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke, confirmed by clinical and radiological evidence
* Ability to understand and follow commands
* willing and able to regularly attend a supervised exercise program

Exclusion Criteria:

* severe cognitive impairment
* Commodity that preclude them from undergoing training and assessment
* Neurological disease other than stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | 6 months
  Functional Independence Measure (FIM) it is an 18-item ordinal scale with seven levels ranging from 1 (total dependence) to 7 (total independence).FIM can be subdivided into a 13-item motor subscale (eating, grooming, bathing, dressing upper body, dressing lower body, personal hygiene, bladder control, bowel control, transfer to tub/shower, walk or wheelchair, stairs) and 5-item cognitive subscale (comprehension, expression, social interaction, problem solving, memory).The motor and cognitive sub-scales scores range from 13 to 91(motor-FIM) and from 5 to 35 (cognitive-FIM). The maximum total score is 126.

SECONDARY OUTCOMES:
motor performance, Fugl-Meyer scale | 6 months
  The Fugl-Meyer physical performance scale assesses five dimensions of impairment, including three aspects of motor control, such as the amplitude of joint movement, pain, sensitivity, motor impairment of the upper and lower extremities and balance. The data are scored in an ordinal scale of 3 (0=no performance; 2=complete performance) applied to each item7. The total motor score is equal to the classification of the upper limb (UL) plus the lower limb (LL), corresponding to 100 total scores (UL=66, LL=34). The total FM score, including the other items, corresponds to 226 scores in the final sum.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, Study Director — Department of Physical therapy,School of Medicine, University of Sao Paulo; Tatiana P Oliveira, Principal Investigator — Department of Physical therapy, School of Medicine, University of Sao Paulo
Locations (1):
- Department of Physical therapy, Medicine School of University of São Paulo, São Paulo, São Paulo, Brazil